CLINICAL TRIAL: NCT06015841
Title: An Adaptive, Phase 2, Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Safety, Tolerability, Immunogenicity, and Pharmacodynamic Effects of ACI-7104.056 in Patients With Early Stages of Parkinson's Disease
Brief Title: A Study to Evaluate the Effects of ACI-7104.056 in Patients With Early Stages of Parkinson's Disease
Acronym: VacSYn
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AC Immune SA (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACI-7104-PD-2103; 2022-500292-31-00 (Other: European Union Clinical Trials Register); 1006102 (Other: Integrated Research Application System)
Record Dates: First submitted 2023-08-04; First posted 2023-08-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Parkinson Disease 6, Early-Onset
Keywords: Early Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Parkinson Disease 6, Autosomal Recessive Early-Onset

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Early PD subjects receive placebo at pre-defined time points over 74 weeks.
  Interventions: Biological: Placebo
- ACI-7104.056 at Dose A (Experimental): Early PD subjects receive dose A of ACI-7104.056 at pre-defined time points over 74 weeks.
  Interventions: Biological: ACI-7104.056 at Dose A
- ACI-7104.056 at Dose B (optional) (Experimental): Early PD subjects receive dose B of ACI-7104.056 at pre-defined time points over 74 weeks. This arm is optional.
  Interventions: Biological: ACI-7104.056 at Dose B (optional)
- ACI-7104.056 at Dose C (optional) (Experimental): Early PD subjects receive dose C of ACI-7104.056 at pre-defined time points over 74 weeks. This arm is optional.
  Interventions: Biological: ACI-7104.056 at Dose C (optional)

INTERVENTIONS:
Biological: Placebo — The placebo is a solution matching the study treatment formulation.
  Arms: Placebo
Biological: ACI-7104.056 at Dose A — The study treatment (ACI-7104.056) consists of an adjuvanted protein peptide conjugate vaccine.
  Arms: ACI-7104.056 at Dose A
Biological: ACI-7104.056 at Dose B (optional) — The study treatment (ACI-7104.056) consists of an adjuvanted protein peptide conjugate vaccine.
  Arms: ACI-7104.056 at Dose B (optional)
Biological: ACI-7104.056 at Dose C (optional) — The study treatment (ACI-7104.056) consists of an adjuvanted protein peptide conjugate vaccine.
  Arms: ACI-7104.056 at Dose C (optional)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, immunogenicity, and pharmacodynamic effects of ACI-7104.056 in patients with early stages of Parkinson's disease.

DETAILED DESCRIPTION:
This is a prospective, multicenter, placebo-controlled, double-blind, randomized study with adaptive features, comprising a screening period of up to 8 weeks, a 74-week double-blind treatment period, and a 26-week post-treatment follow-up period.

Up to 3 cohorts will include 16 subjects each (12 under the study treatment and 4 under placebo; 3:1 active treatment/placebo ratio). One of the initial potential 3 cohorts (Cohorts 2 and 3 are optional) may be expanded in order to reach an overall total of up to 150 subjects in the study. In case a cohort is expanded, the randomization ratio will be adjusted to achieve an active treatment/placebo ratio of 2:1 in this cohort.

The route of administration of the study treatment and placebo will be by intramuscular injections.

ELIGIBILITY:
Inclusion criteria:

1. Confirmed diagnosis of clinically established early PD using the modified Movement Disorder Society criteria, after excluding any other known or suspected cause of PD. The presence of motor symptoms should not be of more than 2 years at screening.
2. Monotherapy treatment with L-Dopa at 300 mg per day, with a stable dose prior to baseline for 3 months. The subject has a reasonably low likelihood of requiring dose adjustment within the next 6 to 12 months after enrolment. Any exception to this rule has to be previously agreed with the Sponsor medical monitor.
3. Male or female.
4. Aged ≥40 to ≤75 years.
5. Body weight range of ≥45 kg to ≤110 kg (99 to 242 lbs) and a body mass index of ≥18 to ≤34 kg/m2.
6. Modified Hoehn-Yahr (H&Y) Stage I to II.
7. A centrally read screening brain DaT-SPECT consistent with PD.
8. Subjects can understand the informed consent form, are able and willing to provide written informed consent, and can be expected to comply with the study protocol according to the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use and local regulations.
9. Female participants must be postmenopausal for at least 1 year and/or surgically sterilized, or, if they are female of childbearing potential or not postmenopausal, they must have a negative blood pregnancy test at screening and be willing to use highly effective methods of contraception from the screening visit until the end of the safety follow-up period (approximately 108 weeks). Male participants in the trial with female partners of childbearing potential are required to use barrier methods of contraception (condoms with spermicide) in addition to contraceptive measures used by female partners during the whole study duration. Men must refrain from donating sperm during this same period. The female partners should use a highly effective method of contraception with a failure rate of less than 1% per year from screening until the end of the safety follow-up period (approximately 108 weeks). The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion criteria:

1. Medical history indicating a Parkinsonian syndrome other than idiopathic PD, including but not limited to, progressive supranuclear palsy, multiple system atrophy, drug induced parkinsonism, essential tremor, vascular parkinsonism, primary dystonia.
2. Known carriers of certain familial PD gene mutations (PRKN, PINK1, DJ1, LRRK2).
3. History of PD-related freezing episodes or falls.
4. History of brain surgery or any neurosurgical procedures.
5. Reside in a nursing home or assisted care facility.
6. A history of cancer within 5 years of baseline with the exception of fully excised non melanoma skin cancers or nonmetastatic prostate cancer that has been stable for at least 6 months, or cervical intraepithelial neoplasia stage I uterine cancer.
7. History of and/or screening brain MRI scan indicative of, clinically significant abnormality including but not limited to prior hemorrhage or infarct >1 cm3 or >3 lacunar infarcts.
8. Diagnosis of a significant central nervous system disease other than PD (including but not limited to Huntington's disease, normal pressure hydrocephalus, cerebrovascular disease including stroke, fronto-temporal dementia, Alzheimer's disease, dementia with Lewy bodies, multiple sclerosis, brain tumor); history of repeated head injury; history of epilepsy or seizure disorder other than febrile seizures as a child.
9. Presence of psychiatric symptoms (eg, confusion, hallucination, delusion, excitation, delirium, abnormal behavior at screening and baseline). Note: mild depression, depressive mood, or mild anxiety arising in the context of PD are not exclusionary.
10. Clinically significant concomitant disease or condition within 6 months prior to screening, or as specified below, that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the study participant:

    1. Autoimmune disease (except well controlled conditions as specified in the study protocol with decision making on a case per case basis).
    2. Any active infectious disease and/or any febrile illness (including noninfectious) within 1 week prior to first dose administration.
    3. Any current psychiatric diagnosis that may interfere with the participant's ability to perform the study.
    4. Women who are pregnant or breastfeeding or intending to become pregnant during the study.
    5. Myocardial infarction within 12 months of baseline.
    6. Known history or documentation of uncontrolled hypotension or bradycardia on more than 1 occasion within 3 months prior to baseline and known history or documentation of uncontrolled hypertension on more than 1 occasion within 3 months prior to baseline (up to Principal Investigator's discretion). Resting pulse rate >100 or <45 bpm. A QT interval corrected using Fridericia's formula measurement of 450 ms for males or 470 ms for females at screening or a family history of long QT-syndrome. Intermittent second or third degree atrioventricular (AV) heart block or AV dissociation or any other clinically significant cardiovascular disease.
    7. Clinically significant abnormalities in laboratory test results at the screening visit (specified in more detail in a separate document), positive result for acute or chronic infectious Hepatitis B virus (HBV; [ie, Hepatitis B surface antigen (HBsAg) positive test]), for Hepatitis C virus (HCV), or for Human Immunodeficiency Virus (HIV) 1 or 2. Successfully treated subjects with HCV (undetectable HCV RNA) are eligible for enrolment. Participants who are immune due to HBV natural infection or HBV vaccination are eligible.
    8. Use of any of the following: monoamine oxidase (MAO)-B inhibitors, catechol-O-methyl transferase (COMT) inhibitors (eg, entacapone, opicapone, tolcapone), amantadine, adenosine A2a antagonists or anticholinergics, or dopaminergic medication (both ergot and nonergot [pramipexole, ropinirole, rotigotine] dopamine agonists) for more than a total of 90 days or within 90 days of baseline.
    9. Antiepileptic medication (eg, valproate) for nonseizure-related treatment that has not remained stable for at least 60 days prior to baseline.
    10. Antidepressant use that has not remained stable for at least 2 months prior to baseline.
    11. Use of any of the following medications within 90 days prior to baseline: metoclopramide, alpha methyldopa, flunarizine, amoxapine, amphetamine derivatives, reserpine, bupropion, buspirone, cocaine, cannabis, mazindol, methamphetamine, methylphenidate, phentermine, phenylpropanolamine, and modafinil. Exceptional use of norephedrine is allowed (eg, treatment for a cold).
    12. Previous participation in a clinical trial using an active immunotherapy against PD, unless there is firm evidence that the subject received placebo only and the placebo formulation is not expected to induce any specific immune response.
    13. Previous treatment with any investigational and/or marketed passive immunotherapy against PD within 6 months before screening or 5 half-lives, whichever is longer, unless there is firm evidence that the subject received placebo only (in the case of any investigational product administered within the frame of a clinical trial participation).
    14. Participation in previous clinical trials for PD and/or for neurological disorders using any small molecule drug with a washout <30 days or <5 half lives of the drug, whichever is longer before screening, unless there is firm evidence that the subject received placebo only.
    15. Concomitant participation in any other clinical trial using experimental or approved medications or therapies (eg, device, stem cell). This does not include noninterventional devices for disease tracking or imaging studies.
    16. Immunomodulating and immunosuppressant drugs including oral corticosteroids within 30 days prior to baseline.
    17. Allergy to any of the components of the study vaccine.
    18. Any contraindications to obtaining a brain MRI or DaT-SPECT, getting a lumbar puncture or receiving IM injections.
11. Current, or history of, alcohol or drug (including cannabis) abuse or other dependence (except nicotine dependence) within 12 months before screening.
12. Subjects with known hypersensitivity to the study vaccine or placebo components.
13. Subjects who previously received a vaccination (ie, influenza vaccine and COVID 19) within the last 4 weeks prior to randomization or standard-of-care immunizations within the last 2 weeks prior to randomization.
14. Subjects being treated with any anticoagulants or antiplatelet drugs, except aspirin at doses of 100 mg daily or lower.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) assessed by intensity (mild, moderate or severe) and causal relationship (unrelated, or unlikely, possibly, probably or definitely related) | From Screening (ICF signature) to Week 100
Number of participants with abnormal MRI results | From Baseline to Week 100
Number of participants with clinically significant changes in physical and neurological examination results | From Baseline to Week 74
Number of participants reporting suicidal ideation or behavior using Columbia-Suicide Severity Rating Scale (C-SSRS) | From Baseline to Week 100
Measurement of levels of specific antibodies against a-synuclein present in serum generated by ACI-7104.056 | From Baseline to Week 100

SECONDARY OUTCOMES:
Measures of alpha-synuclein (a-syn) related biofluid biomarkers | From Baseline to Week 100
Measurement of levels of dopamine transporter proteins in specific brain regions, notably substantia nigra, by Dopamine Transporter-Single Photon Emission Computerized Tomography (DaT-SPECT) imaging | From Baseline to Week 100
Change from baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III | From Baseline to Week 100

OTHER OUTCOMES:
Change in motor and nonmotor functions using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | From Baseline to Week 100

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Berg, Prof., Study Chair — Klinik für Neurologie, UKSH Campus Kiel, Germany
Locations (12):
- Germany (3):
  - Katholisches Klinikum Bochum GmbH, Bochum
  - Paracelsus-Kliniken Deutschland GmbH & Co. KGaA, Kassel
  - University Medical Centre Schleswig-Holstein, Kiel
- Spain (6):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Policlinica Gipuzkoa, Donostia / San Sebastian
  - Hospital Universitario De La Princesa, Madrid
  - Hospital Universitario Puerta De Hierro De Majadahonda, Majadahonda
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
- United Kingdom (3):
  - King's College Hospital NHS Foundation Trust, London
  - Re:Cognition Health Limited, London
  - Northern Care Alliance NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Volc D, Poewe W, Kutzelnigg A, Luhrs P, Thun-Hohenstein C, Schneeberger A, Galabova G, Majbour N, Vaikath N, El-Agnaf O, Winter D, Mihailovska E, Mairhofer A, Schwenke C, Staffler G, Medori R. Safety and immunogenicity of the alpha-synuclein active immunotherapeutic PD01A in patients with Parkinson's disease: a randomised, single-blinded, phase 1 trial. Lancet Neurol. 2020 Jul;19(7):591-600. doi: 10.1016/S1474-4422(20)30136-8. PMID 32562684